CLINICAL TRIAL: NCT00786513
Title: Randomized Double Blind Controlled Trial of the Use of a Biofilm Antimicrobial Susceptibility Assay to Guide Antibiotic Therapy in Chronic Pseudomonas Aeruginosa Infected Cystic Fibrosis Patients
Brief Title: Use of a Biofilm Antimicrobial Susceptibility Assay to Guide Antibiotic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Valerie Waters, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000011132
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Pseudomonas aeruginosa; biofilm; antibiotic susceptibility testing; pediatrics
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Other: Conventional antimicrobial susceptibility testing
- Intervention Arm (Experimental)
  Interventions: Other: Biofilm antimicrobial susceptibility testing

INTERVENTIONS:
Other: Conventional antimicrobial susceptibility testing — Subjects in this arm will be prescribed 14 days of an intravenous 2 drug antibiotic combination based on conventional planktonic antimicrobial susceptibility testing results.
  Arms: Control Arm
Other: Biofilm antimicrobial susceptibility testing — Subjects in this arm will be prescribed 14 days of an intravenous 2 drug antibiotic combination based on biofilm antimicrobial susceptibility testing results.
  Arms: Intervention Arm

SUMMARY:
The purpose of this study is to determine whether choosing antibiotics based on a biofilm antimicrobial susceptibility assay rather than a conventional planktonic antimicrobial susceptibility assay to treat CF patients with chronic P. aeruginosa infection with an acute pulmonary exacerbation is a safe intervention that will result in improved microbiological and clinical outcomes and decrease markers of pulmonary inflammation.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common fatal genetic condition in the Caucasian population and affects over 3,000 Canadians. Respiratory failure caused by chronic pulmonary infection is the primary cause of death in CF patients. The improved life expectancy of CF patients in the past several decades is due in part to the more aggressive use of antibiotics in the treatment of respiratory infections. However, there is currently no antimicrobial susceptibility assay that can predict which antibiotics will result in improved patient outcomes. Since Pseudomonas aeruginosa is known to grow as a resistant biofilm in the CF lung, antimicrobial susceptibility testing based on biofilm growth of P. aeruginosa may lead to different antibiotic choices that significantly decrease the pulmonary bacterial density of P. aeruginosa. A biofilm antimicrobial susceptibility assay thus has the ability to change the way antibiotics are chosen to treat CF patients and result in improved lung function and longer lives for all CF patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on the following: sweat chloride > 60 mEq/L or genotype with 2 identifiable mutations consistent with CF; and one or more clinical features consistent with CF
* Chronically infected with P. aeruginosa (>50% of respiratory specimens positive for P. aeruginosa in the 24 months prior to screening)
* Able to produce sputum (expectorated or induced)
* Able to reproducibility perform pulmonary function testing
* Written informed consent provided

Exclusion Criteria:

* Sputum culture negative for P. aeruginosa or with a density of less that 10^5 CFU/g at screening
* Sputum culture positive for Burkholderia cepacia at screening
* History of B. cepacia positive respiratory culture within 24 months prior to screening
* Use of antibiotics other than those prescribed by the principal investigator
* History of allergy (urticarial rash, diffuse erythroderma, serum sickness) to more than two groups of antibiotics (aminoglycosides, penicillins, cephalosporins, monobactams, macrolides, or quinolones) that are a therapeutic option
* History of anaphylaxis or other life threatening complication to any antibiotic in the six groups that are a therapeutic option
* Post lung transplantation or listed for lung transplantation
* Pregnancy
* A septic or clinically unstable patient
* Presence of a condition or abnormality that in the opinion of an investigator would compromise the safety of the patient or the quality of the data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in the intervention arm versus the control arm who have ≥ 3 log drop in colony forming units (CFUs) of P. aeruginosa in sputum. | Measured at day 0 and day 14 of antibiotic treatment and at the 1 month follow-up visit

SECONDARY OUTCOMES:
The change in pulmonary function tests, including forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and maximal midexpiratory flow rate (FEF25-75) in the intervention arm versus the control arm | Measured at day 0, day 7, and day 14 of antibiotic treatment and at the 1 month follow-up visit
The time to subsequent acute pulmonary exacerbation in the intervention arm versus the control arm | 1 year following the completion of antibiotic therapy
The change in the cumulative score on a quality of life questionnaire in the intervention arm versus the control arm | Measued at day 0 and day 14 of antibiotic treatment and at the 1 month follow-up visit
The change in the measurement of markers of pulmonary inflammation (neutrophil counts, neutrophil elastase and IL-8 levels in sputum) in the intervention arm versus the control arm. | Meaured at day 0 and day 14 of antibiotic treatment and at the 1 month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Waters, MD, Principal Investigator — The Hospital for Sick Children; Yvonne Yau, MD, Principal Investigator — The Hospital for Sick Children
Locations (5):
- Canada (5):
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Yau YC, Ratjen F, Tullis E, Wilcox P, Freitag A, Chilvers M, Grasemann H, Zlosnik J, Speert D, Corey M, Stanojevic S, Matukas L, Leahy TR, Shih S, Waters V. Randomized controlled trial of biofilm antimicrobial susceptibility testing in cystic fibrosis patients. J Cyst Fibros. 2015 Mar;14(2):262-6. doi: 10.1016/j.jcf.2014.09.013. Epub 2014 Oct 30. PMID 25453872